CLINICAL TRIAL: NCT05849714
Title: Validation Study of a Peri-intervention Diabetes Management Algorithm (DIAPI) for Endoscopy Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2023-11359
Record Dates: First submitted 2023-04-25; First posted 2023-05-09 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus
Keywords: Peri-procedural; Endoscopy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Patients will receive usual care for their diabetes during their peri-procedural period.
  Interventions: Other: Usual Care
- DIAPI (Experimental): Patients will receive the care for their diabetes recommended by the DIAPI algorithm during their peri-procedural period.
  Interventions: Other: Peri-intervention Diabetes Management Algorithm (DIAPI)

INTERVENTIONS:
Other: Peri-intervention Diabetes Management Algorithm (DIAPI) — Patients and healthcare workers will apply DIAPI's orders.
  Arms: DIAPI
Other: Usual Care — Patients and healthcare workers will apply the mainstay management, which is using the treating-physician's recommendations instead of DIAPI's.
  Arms: Usual Care

SUMMARY:
The peri-endoscopy management of diabetes mellitus creates significant challenges for both patients and healthcare professionals. These procedures require fasting and in certain situations, such as prior to a colonoscopy, the diet must be modified the day before the intervention and patients need to take a laxative. These factors put patients at high risk for hyperglycemia and hypoglycemia. Inadequate diabetes control or the continuation of certain medications during this period can be dangerous for the patient and lead to the cancellation of the procedure.

DIAPI is a web application designed to generate orders for optimal and personalized treatment based on each patient's antidiabetic treatment, their glycemic control, their risk of hypoglycemia, and the intervention-related variables. DIAPI's algorithm is established on current evidence-based data when available, and experts' opinions.

Information generated by DIAPI:

* For the patient: Clear instructions regarding their diabetes medication management for the days preceding and the day of the endoscopy.
* For the health care team:

  * Clear instructions regarding patient's diabetes medication management for the days preceding and the day of the endoscopy;
  * Individualized hyperglycemia protocol;
  * Hypoglycemia protocol;
  * Guidelines if SGLT2 inhibitors have not been discontinued pre-intervention;
  * Suggestion on whether an Endocrinology consultation is needed.

DIAPI aims to simplify the complex task of peri-intervention diabetes management while ensuring patient safety. It is a cost-effective solution that can lead to a reduction of unnecessary Endocrinology consultations, a decrease in nurses' workload, a lessening of the risk of errors and a diminution of endoscopy cancellation.

The validation study is divided into two main phases.

* Phase 1 - Concordance. The investigators will assess the reproducibility of DIAPI orders when two different healthcare workers (an endocrinologist and a nurse) collect data for the same patient. The investigators hypothesize that DIAPI orders are concordant in 80%. Patients in this phase will be subjected to the mainstay management, which is using the treating-physician's recommendations instead of DIAPI's. This group will be the control arm for the non-inferiority study (Phase 2).
* Phase 2 - Non-inferiority study. The investigators hypothesize that DIAPI's orders are not inferior to the recommendations issued by the treating-physician in terms of efficacy and security. Patients in this phase will be subjected DIAPI's orders. This group will be the intervention arm for the non-inferiority study.

ELIGIBILITY:
Inclusion Criteria:

* Living with diabetes mellitus for at least 6 months
* Receiving pharmacological treatment for diabetes mellitus
* Awaiting an endoscopy intervention scheduled in 2 weeks or more in order to have time to prepare for the study participation

Exclusion Criteria:

* Undergoing an urgent endoscopy intervention
* Being pregnant
* Currently treated with an insulin pump or the insulin Entuzity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Concordance rate of duplicate prescriptions generated by DIAPI when two different healthcare workers collect data for the same patient. (Part 1 of study) | 1 week
  Concordance and discordance are dichotomic concepts. To classify this binary issue, the investigators use a home-made ''Difference Score''. The components of this score have been established to ensure patient safety by minimizing the risk of hypoglycemia, hyperglycemia, and diabetic ketoacidosis.
  * Concordance = difference score of ≤ 25.0 %.
  * Discordant= difference score of > 25.0 %.
proportion of patients with glycaemia level within target from arrival to departure from the endoscopy unit, i.e. between 4 - 10 mmol/L. (Part 2 of study) | 1 day
  The glycaemia will be measured at least every hour for the duration of the stay in the endoscopy unit.

SECONDARY OUTCOMES:
Proportion of DIAPI orders for which the endocrinologist disagrees with at least one of its recommendations. (Part 1 of study) | 1 week
Proportion of participants for whom an endocrinology consultation was recommended by DIAPI. (Part 1 of study) | 1 week
Healthcare workers' satisfaction level with the use of DIAPI, assessed by a questionnaire. (Part 1 of study) | 1 week
Proportion of participants who followed DIAPI recommendations. (Part 2 of study) | 1 week
• Proportion of canceled endoscopies due to dysglycemia, ketoacidosis or for reasons related to diabetes management. (Part 2 of study) | 1 week
Proportion of participants hospitalized for a diabetes-related condition. (Part 2 of study) | 1 month
Proportion of participants who experienced: episode of hypoglycemia <3 and < 4 mmol/L, episode of hyperglycemia >10, > 15 and >20 mmol/L, episode of ketoacidosis. (Part 2 of study) | 1 week
  These episodes will be reported by time frame: the day before, the same day and the day after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marie Boutin, MD, PhD, Principal Investigator — Université de Montréal
Locations (1):
- Centre hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No